CLINICAL TRIAL: NCT00032136
Title: An Open Label, Randomized Multicenter Comparative Trial Of 5 Years Adjuvant Exemestane Treatment Versus 5 Years Adjuvant Tamoxifen Treatment In Postmenopausal Women With Early Breast Cancer
Brief Title: Exemestane Compared With Tamoxifen in Treating Postmenopausal Women With Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cancer Research Campaign Clinical Trials Centre (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CRC-TU-TEAM; CDR0000069260 (Registry Identifier: PDQ (Physician Data Query)); EU-20149; ISRCTN75225940
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2007-03

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane; Tamoxifen; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: exemestane
Drug: tamoxifen citrate
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of breast cancer cells. Hormone therapy using exemestane may fight breast cancer by reducing the production of estrogen. It is not yet known if exemestane is more effective than tamoxifen in preventing the recurrence of breast cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of exemestane with that of tamoxifen in treating postmenopausal women who have undergone surgery to remove early-stage breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy and tolerability of adjuvant exemestane versus adjuvant tamoxifen in postmenopausal women with early breast cancer.
* Compare the relapse-free survival and overall survival of patients treated with these drugs.
* Compare the incidence of contralateral breast cancer in patients treated with these drugs.
* Compare the safety and long-term tolerability of these drugs in these patients.
* Compare the quality of life of patients treated with these drugs.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to estrogen receptor (ER)/progesterone receptor (PgR) status (ER positive vs ER negative/PgR positive vs ER positive/PgR unknown), prior chemotherapy (none vs taxane-based vs anthracycline-based vs other), and nodal status (negative vs 1-3 nodes positive vs 4 or more nodes positive). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral tamoxifen once daily
* Arm II: Patients receive oral exemestane once daily. Treatment in both arms continues for a minimum of 5 years in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline and at months 3 and 12 during study.

Patients are followed at least annually.

PROJECTED ACCRUAL: Approximately 4,400 patients (2,200 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed early adenocarcinoma of the breast

  * Completely excised by surgery with curative intent (R0)

    * Any N OR
    * Any primary tumor greater than 3 cm OR
    * Any primary tumor grade III and greater than 1 cm
  * M0
* No positive supraclavicular nodes
* Hormone receptor status:

  * Estrogen and/or progesterone receptor positive

PATIENT CHARACTERISTICS:

Age:

* Any age
* See Menopausal status

Sex:

* Female

Menopausal status:

* Postmenopausal

  * Any age with bilateral oophorectomy or amenorrhea for at least 5 years OR
  * Age 50 or over:

    * Natural amenorrhea for at least 1 year OR
    * Chemotherapy-induced amenorrhea for at least 2 years OR
    * Radiation-induced amenorrhea (at least 3 months since prior radiotherapy) OR
  * Under age 50:

    * If amenorrheic for less than 5 years (any cause) or prior hysterectomy without bilateral surgical oophorectomy, follicle-stimulating hormone must be assayed to confirm postmenopausal status

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Platelet count greater than 100,000/mm3
* WBC greater than 3,000/mm3

Hepatic:

* SGOT or SGPT less than 2.5 times upper limit of normal (ULN)

Renal:

* Creatinine less than 1.5 times ULN

Cardiovascular:

* No uncontrolled cardiac disease
* No unstable angina
* No congestive heart failure or arrhythmia requiring medical therapy
* No myocardial infarction within the past 3 months

Other:

* No severe osteoporosis
* No other malignancies within the past 5 years except adequately treated carcinoma in situ of the cervix or basal cell skin cancer
* No other serious concurrent disease that would preclude study
* No psychiatric disorders that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior neoadjuvant chemotherapy
* No more than 10 weeks since completion of prior adjuvant chemotherapy

Endocrine therapy:

* No prior adjuvant hormonal therapy for breast cancer
* No prior neoadjuvant hormonal therapy (prior to surgery) for duration of more than 4 weeks
* At least 4 weeks since prior hormone replacement therapy

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics
* No more than 10 weeks since completion of curative surgery

Other:

* No other concurrent investigational agents or participation in another clinical study (except adjuvant cytotoxic chemotherapy studies)
* Concurrent bisphosphonates allowed

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4400 (Estimated)
Dates: Start 2001-12; Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Relapse-free survival

SECONDARY OUTCOMES:
Overall survival
Incidence of second breast cancer in contralateral breast
Safety and long term tolerability
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rea, MD, Study Chair — City Hospital Birmingham
Locations (1):
- City Hospital - Birmingham, Birmingham, England, United Kingdom

REFERENCES:
- [Background] Hadji P, Asmar L, van Nes JG, Menschik T, Hasenburg A, Kuck J, Nortier JW, van de Velde CJ, Jones SE, Ziller M. The effect of exemestane and tamoxifen on bone health within the Tamoxifen Exemestane Adjuvant Multinational (TEAM) trial: a meta-analysis of the US, German, Netherlands, and Belgium sub-studies. J Cancer Res Clin Oncol. 2011 Jun;137(6):1015-25. doi: 10.1007/s00432-010-0964-y. Epub 2010 Dec 18. PMID 21170551
- [Result] van de Velde CJ, Rea D, Seynaeve C, Putter H, Hasenburg A, Vannetzel JM, Paridaens R, Markopoulos C, Hozumi Y, Hille ET, Kieback DG, Asmar L, Smeets J, Nortier JW, Hadji P, Bartlett JM, Jones SE. Adjuvant tamoxifen and exemestane in early breast cancer (TEAM): a randomised phase 3 trial. Lancet. 2011 Jan 22;377(9762):321-31. doi: 10.1016/S0140-6736(10)62312-4. PMID 21247627
- [Result] Kieback DG, Harbeck N, Bauer W, Hadji P, Weyer G, Menschik T, Hasenburg A. Endometrial effects of exemestane compared to tamoxifen within the Tamoxifen Exemestane Adjuvant Multicenter (TEAM) trial: results of a prospective gynecological ultrasound substudy. Gynecol Oncol. 2010 Dec;119(3):500-5. doi: 10.1016/j.ygyno.2010.08.006. Epub 2010 Sep 15. PMID 20832103
- [Result] Hadji P, Ziller M, Kieback DG, Dornoff W, Tessen HW, Menschik T, Kuck J, Melchert F, Hasenburg A. Effects of exemestane and tamoxifen on bone health within the Tamoxifen Exemestane Adjuvant Multicentre (TEAM) trial: results of a German, 12-month, prospective, randomised substudy. Ann Oncol. 2009 Jul;20(7):1203-9. doi: 10.1093/annonc/mdn762. Epub 2009 Feb 13. PMID 19218306
- [Result] Hadji P, Ziller M, Kieback DG, Menschik T, Kalder M, Kuck J, Hasenburg A. The effect of exemestane or tamoxifen on markers of bone turnover: results of a German sub-study of the Tamoxifen Exemestane Adjuvant Multicentre (TEAM) trial. Breast. 2009 Jun;18(3):159-64. doi: 10.1016/j.breast.2009.03.003. Epub 2009 Apr 11. PMID 19364653
- [Derived] Leblanc A, Beltran-Bless AA, Pond GR, El Emam K, Juwara L, Clemons L, Bayani J, Pilgram L, Pharoah P, Mallon E, Taylor KJ, Markopoulos C, Dirix L, Vandermeer L, Hilton J, Savard MF, Bartlett JMS, Clemons M. Prognostic and predictive performance of PREDICT 2.1, PREDICT v3, and RSClin in node-negative early breast cancer: a TEAM pathology substudy. Breast Cancer Res Treat. 2026 Feb 5;215(3):74. doi: 10.1007/s10549-026-07909-5. PMID 41642493
- [Derived] Beltran-Bless AA, Pond GR, Bayani J, Barker SL, Spears M, Mallon E, Taylor KJ, Hasenburg A, Markopoulos C, Dirix L, Meershoek-Klein Kranenbarg E, van de Velde CJH, Rea DW, Vandermeer L, Hilton J, Bartlett JMS, Clemons M. Does RSClin provide additional information over classic clinico-pathologic scores (PREDICT 2.1, INFLUENCE 2.0, CTS5)? Breast. 2025 Oct;83:104528. doi: 10.1016/j.breast.2025.104528. Epub 2025 Jul 4. PMID 40633461
- [Derived] Bayani J, Kornaga EN, Crozier C, Jang GH, Bathurst L, Kalatskaya I, Trinh QM, Yao CQ, Livingstone J, Boutros PC, Spears M, McPherson JD, Stein LD, Rea D, Bartlett JMS. Identification of Distinct Prognostic Groups: Implications for Patient Selection to Targeted Therapies Among Anti-Endocrine Therapy-Resistant Early Breast Cancers. JCO Precis Oncol. 2019 Dec;3:1-13. doi: 10.1200/PO.18.00373. PMID 35100692
- [Derived] Derks MGM, Bastiaannet E, van de Water W, de Glas NA, Seynaeve C, Putter H, Nortier JWR, Rea D, Hasenburg A, Markopoulos C, Dirix LY, Portielje JEA, van de Velde CJH, Liefers GJ. Impact of age on breast cancer mortality and competing causes of death at 10 years follow-up in the adjuvant TEAM trial. Eur J Cancer. 2018 Aug;99:1-8. doi: 10.1016/j.ejca.2018.04.009. Epub 2018 Jun 6. PMID 29885375
- [Derived] Derks MGM, Blok EJ, Seynaeve C, Nortier JWR, Kranenbarg EM, Liefers GJ, Putter H, Kroep JR, Rea D, Hasenburg A, Markopoulos C, Paridaens R, Smeets JBE, Dirix LY, van de Velde CJH. Adjuvant tamoxifen and exemestane in women with postmenopausal early breast cancer (TEAM): 10-year follow-up of a multicentre, open-label, randomised, phase 3 trial. Lancet Oncol. 2017 Sep;18(9):1211-1220. doi: 10.1016/S1470-2045(17)30419-9. Epub 2017 Jul 18. PMID 28732650
- [Derived] Bartlett JM, Brookes CL, Piper T, van de Velde CJ, Stocken D, Lyttle N, Hasenburg A, Quintayo MA, Kieback DG, Putter H, Markopoulos C, Kranenbarg EM, Mallon EA, Dirix LY, Seynaeve C, Rea DW. Do type 1 receptor tyrosine kinases inform treatment choice? A prospectively planned analysis of the TEAM trial. Br J Cancer. 2013 Oct 29;109(9):2453-61. doi: 10.1038/bjc.2013.609. Epub 2013 Oct 3. PMID 24091623